CLINICAL TRIAL: NCT06009237
Title: A Study to Evaluate Pharmacokinetics, Safety, and Tolerability of ABBV-903 in Healthy Japanese and Han Chinese Subjects
Brief Title: A Study to Assess Pharmacokinetics, Safety, and Tolerability of ABBV-903 in Healthy Japanese and Han Chinese Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: M24-227
Record Dates: First submitted 2023-08-21; First posted 2023-08-24 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Healthy Volunteers
Keywords: ABBV-903; Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Part 1: Han-Chinese Participants ABBV-903 (Experimental): Han-Chinese participants will receive a single dose of ABBV-903.
  Interventions: Drug: ABBV-903
- Part 1: Japanese Participants ABBV-903 (Experimental): Japanese participants will receive a single dose of ABBV-903.
  Interventions: Drug: ABBV-903
- Part 1: Placebo (Experimental): Participants will receive a single dose of Placebo for ABBV-903.
  Interventions: Drug: Placebo for ABBV-903
- Part 2: Japanese Participants ABBV-903 (Experimental): Japanese participants will receive ABBV-903 daily for 10 days.
  Interventions: Drug: ABBV-903
- Part 2: Japanese Participants Placebo (Experimental): Japanese participants will receive placebo daily for 10 days.
  Interventions: Drug: Placebo for ABBV-903

INTERVENTIONS:
Drug: ABBV-903 — Tablet; oral
  Arms: Part 1: Han-Chinese Participants ABBV-903; Part 1: Japanese Participants ABBV-903; Part 2: Japanese Participants ABBV-903
Drug: Placebo for ABBV-903 — Tablet; oral
  Arms: Part 1: Placebo; Part 2: Japanese Participants Placebo

SUMMARY:
The objective of this study is to assess the pharmacokinetics (PK), safety, and tolerability of ABBV-903 or placebo in healthy adult Japanese and Han Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

- Healthy Japanese or Han Chinese male or female; age is between 18 and 65 years, inclusive at the time of screening.

* Han Chinese subject must be first-generation Han Chinese of full Chinese parentage residing outside of China. Subjects must maintain a typical Chinese lifestyle, including consuming a typical Chinese diet.

OR

* Japanese subject must be first- or second generation Japanese of full Japanese parentage. First-generation subjects will have been born in Japan to two parents and four grandparents also born in Japan of full Japanese descent. Second-generation subjects born outside of Japan must have two parents and four grandparents born in Japan of full Japanese descent. All subjects must maintain a typical Japanese lifestyle, including consuming a typical Japanese diet.

  * Body Mass Index (BMI) is >= 18.0 to <= 30.0 kg/m2 after rounding to the tenths decimal, at screening and upon initial confinement. BMI is calculated as weight in kg divided by the square of height measured in meters.

Exclusion Criteria:

* History of any clinically significant illness/infection/major febrile illness, hospitalization, as determined by the investigator, or any surgical procedure within 30 days prior to the first dose of study drug.
* Evidence of dysplasia or history of malignancy (including lymphoma and leukemia) other than successfully treated non-metastatic cutaneous squamous cell, basal cell carcinoma orlocalized carcinoma in situ of the cervix.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of ABBV-903 | Up to Day 4
  Cmax of ABBV-903 will be assessed.
Time to Cmax (Tmax) of ABBV-903 | Up to Day 4
  Tmax of ABBV-903 will be assessed.
Apparent Terminal Phase Elimination Rate Constant (β) of ABBV-903 | Up to Day 4
  Apparent terminal phase elimination rate constant (β) of ABBV-903 will be assessed.
Terminal Phase Elimination Half-life (t1/2) of ABBV-903 | Up to Day 4
  Terminal phase elimination half-life (t1/2) of ABBV-903 will be assessed.
Area under the Plasma Concentration-time Curve (AUC) from Time 0 to the Time t (AUC0-t) of ABBV-903 | Up to Day 4
  AUC0-t of ABBV-903 will be assessed.
AUC from Time 0 to Infinity (AUC0-inf) of ABBV-903 | Up to Day 4
  AUC0-inf of ABBV-903 will be assessed.
Number of Participants with Adverse Events (AEs) | Baseline to Day 34
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Anaheim Clinical Trials LLC /ID# 257033, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No